CLINICAL TRIAL: NCT07267039
Title: Comparison of Phenol Neurolysis and Local Anesthetic Plus Steroid Genicular Nerve Block Under Ultrasound Guidance in Patients With Knee Osteoarthritis: Effects on Pain, Function, and Safety
Brief Title: Phenol Neurolysis Versus Local Anesthetic Plus Steroid Genicular Nerve Block in Knee Osteoarthritis
Status: Active, not recruiting | Type: Observational
Sponsor: Salim Sencar (Other)
Responsible Party: Sponsor-Investigator, Salim Sencar, Resident Physician (Research Assistant), Department of Physical Medicine and Rehabilitation, Ondokuz Mayıs University Faculty of Medicine, Ondokuz Mayıs University
Organization: Ondokuz Mayıs University (Other)
Other Study IDs: OMU-FTR-2025/44; OMU-EC-2025-44 (Other: Ondokuz Mayıs University Clinical Research Ethics Committee)
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-10

CONDITIONS: Knee Osteoarthritis; Genicular Nerve Block
Keywords: Knee Osteoarthritis; Gonarthrosis; Genicular Nerve Block; Genicular Nerve Neurolysis; Phenol; Bupivacaine; Triamcinolone Acetonide
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Phenol; Bupivacaine; Triamcinolone Acetonide; Anesthetics, Local

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Phenol Neurolysis: Patients in this group receive ultrasound-guided genicular nerve neurolysis. Using a 22G, 50 mm needle under ultrasound guidance, injections are performed at the superomedial, superolateral, and inferomedial genicular nerves. At each site, 2 mL of 6% phenol is injected to achieve chemical neurolysis and long-term pain relief.
  Interventions: Drug: Phenol Injection
- Local Anesthetic + Triamcinolone Acetonide Block: Patients in this group receive ultrasound-guided genicular nerve block. At the same three target nerves (superomedial, superolateral, inferomedial), 2 mL of a mixture containing 0.25% bupivacaine and 20 mg triamcinolone acetonide is injected at each site. This combination provides nerve blockade with additional anti-inflammatory effect from the corticosteroid.
  Interventions: Drug: Bupivacaine + Triamcinolone Acetonide Injection

INTERVENTIONS:
Drug: Phenol Injection — Ultrasound-guided genicular nerve neurolysis performed at the superomedial, superolateral, and inferomedial genicular nerves. A 22G, 50 mm insulated needle is placed under ultrasound guidance, and 2 mL of 6% phenol is injected at each target site for chemical neurolysis.
  Other Names: Phenol Neurolysis
  Groups: Phenol Neurolysis
Drug: Bupivacaine + Triamcinolone Acetonide Injection — Ultrasound-guided genicular nerve block performed at the superomedial, superolateral, and inferomedial genicular nerves. At each site, 2 mL of a solution containing 0.25% bupivacaine and 20 mg triamcinolone acetonide is injected using a 22G, 50 mm insulated needle. This provides both local anesthetic and anti-inflammatory effects.
  Other Names: Local Anesthetic + Steroid Block
  Groups: Local Anesthetic + Triamcinolone Acetonide Block

SUMMARY:
This study aims to evaluate two different ultrasound-guided procedures for patients with knee osteoarthritis (gonarthrosis) who did not benefit from conservative treatments. The first method is genicular nerve neurolysis with phenol, a chemical agent that blocks nerve signals and may reduce pain for a longer period. The second method is a genicular nerve block with local anesthetic (bupivacaine) and corticosteroid (triamcinolone acetonide), which is commonly used to relieve pain and inflammation.

A total of 42 patients are followed prospectively. Pain intensity is measured using the Visual Analog Scale (VAS), and functional outcomes are assessed with the WOMAC Index and Oxford Knee Score (OKS). Joint range of motion, need for pain medications, and possible side effects are also monitored.

The results will help to compare the effectiveness and safety of phenol neurolysis and triamcinolone acetonide-local anesthetic nerve block, and may guide future treatment choices for patients with knee osteoarthritis.

DETAILED DESCRIPTION:
Knee osteoarthritis (gonarthrosis) is a major cause of chronic pain and disability. Patients who fail to respond to conservative treatments such as medications, physical therapy, and exercise often require interventional options for pain relief.

This prospective observational cohort study compares two ultrasound-guided procedures targeting the genicular nerves of the knee:

Genicular nerve neurolysis with phenol - phenol induces protein denaturation and Wallerian degeneration in nerve fibers, providing long-term analgesia.

Genicular nerve block with local anesthetic (bupivacaine) and corticosteroid (triamcinolone acetonide) - this combination offers immediate pain reduction from nerve blockade and potential prolonged relief due to the anti-inflammatory action of the steroid.

A total of 42 patients with Kellgren-Lawrence grade 3-4 knee osteoarthritis and moderate-to-severe pain (VAS ≥ 4 for ≥ 3 months) are prospectively followed. Interventions are performed under ultrasound guidance at the superomedial, superolateral, and inferomedial genicular nerves.

The primary outcome is change in pain severity (VAS). Secondary outcomes include functional improvement assessed by the WOMAC Index and Oxford Knee Score (OKS), joint range of motion, need for nonsteroidal anti-inflammatory drugs (NSAIDs), and procedure-related adverse events. Assessments are performed at baseline, 2 weeks, and 3 months post-procedure.

The study aims to provide comparative evidence on the effectiveness and safety of phenol neurolysis versus triamcinolone acetonide-local anesthetic block, helping to guide clinical practice in the management of knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 years
* Diagnosis of knee osteoarthritis (Kellgren-Lawrence grade 3-4) confirmed by radiographic evaluation
* Moderate to severe knee pain for at least 3 months (VAS ≥ 4)
* Inadequate response to conservative treatments (e.g., medications, physical therapy, exercise)
* Ability to provide informed consent

Exclusion Criteria:

* History of knee surgery (e.g., total knee arthroplasty) on the affected side
* Intra-articular injection (hyaluronic acid, corticosteroid, PRP, etc.) within the last 6 months
* Secondary arthritis (e.g., rheumatoid arthritis, gout, septic arthritis, trauma-related arthritis)
* Severe coagulopathy or current use of anticoagulant therapy contraindicating injection
* Local skin infection at the injection site
* Known allergy or contraindication to phenol, bupivacaine, or triamcinolone acetonide
* Severe uncontrolled systemic disease (e.g., advanced cardiac, hepatic, or renal failure)
* Pregnancy or breastfeeding

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients (≥40 years) diagnosed with moderate to severe knee osteoarthritis (Kellgren-Lawrence grade 3-4) who did not benefit from conservative treatments such as medications and physical therapy. A total of 42 patients are enrolled and treated at the Physical Medicine and Rehabilitation Department, Ondokuz Mayis University, Faculty of Medicine, Samsun, Turkey.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Intensity Measured by Visual Analog Scale (VAS) | Baseline, 2 weeks, and 3 months after the intervention
  Pain severity will be evaluated using the Visual Analog Scale (VAS; 0-10 cm), where 0 indicates no pain and 10 indicates the worst imaginable pain. Patients will rate their knee pain at rest and during activity. The main outcome is the change in VAS score from baseline to follow-up assessments.

SECONDARY OUTCOMES:
Change in Function and Symptoms Measured by Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Baseline, 2 weeks, 3 months, and 6 months after the intervention
  The WOMAC Index will be used to assess three domains: pain, stiffness, and physical function in patients with knee osteoarthritis. Scores will be calculated according to the standard WOMAC scoring system, with higher scores indicating worse symptoms. The outcome is the change in WOMAC score from baseline to follow-up.
Change in Knee Function Measured by Oxford Knee Score (OKS) | Baseline, 2 weeks, 3 months, and 6 months after the intervention
  he Oxford Knee Score (OKS) is a 12-item patient-reported outcome measure evaluating pain and physical function related to the knee. Scores range from 0 to 48, with higher scores indicating better function. The outcome is the change in OKS from baseline to follow-up.
Change in Knee Range of Motion (ROM) | Baseline, 2 weeks, 3 months, and 6 months after the intervention
  Knee joint range of motion, including flexion and extension, will be measured using a goniometer by a blinded assessor. Both active and passive ROM will be recorded. The outcome is the change in degrees of movement compared to baseline.
Change in Nonsteroidal Anti-inflammatory Drug (NSAID) Consumption | Baseline to 2 weeks, 2 weeks to 3 months, and 3 to 6 months after the intervention
  The number of NSAID doses consumed by participants will be recorded throughout the follow-up period. The outcome measure is the total NSAID use and change compared to baseline.
Adverse Events Related to the Intervention | Baseline through 6 months after the intervention
  Any adverse events possibly or probably related to the intervention will be recorded, including local complications (infection, bleeding, hematoma, skin changes) or systemic side effects.

CONTACTS AND LOCATIONS:
Overall Officials: Bora UZUNER, MD (Medical Doctor), Principal Investigator — Ondokuz Mayis University, Faculty of Medicine, Department of Physical Medicine and Rehabilitation; Salim SENCAR, MD (Medical Doctor), Study Director — Ondokuz Mayis University, Faculty of Medicine, Department of Physical Medicine and Rehabilitation
Locations (1):
- Ondokuz Mayis University, Faculty of Medicine, Department of Physical Medicine and Rehabilitation, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because this is a single-center thesis study with a small number of patients, and data are not intended for public repositories. Only aggregated, anonymized results will be published.

REFERENCES:
- [Result] Risso RC, Ferraro LHC, Nouer Frederico T, Peng PWH, Luzo MV, Debieux P, Sakata RK. Chemical Ablation of Genicular Nerve with Phenol for Pain Relief in Patients with Knee Osteoarthritis: A Prospective Study. Pain Pract. 2021 Apr;21(4):438-444. doi: 10.1111/papr.12972. Epub 2020 Dec 29. PMID 33277760
- [Result] Shanahan EM, Robinson L, Lyne S, Woodman R, Cai F, Dissanayake K, Paddick K, Cheung G, Voyvodic F. Genicular Nerve Block for Pain Management in Patients With Knee Osteoarthritis: A Randomized Placebo-Controlled Trial. Arthritis Rheumatol. 2023 Feb;75(2):201-209. doi: 10.1002/art.42384. Epub 2022 Nov 11. PMID 36369781
- See also: American College of Rheumatology (ACR) Guideline for the Management of Osteoarthritis of the Knee — https://rheumatology.org
- See also: National Institute for Health and Care Excellence (NICE) Guideline for Osteoarthritis: Care and Management — https://www.nice.org.uk/guidance/cg177